CLINICAL TRIAL: NCT03919916
Title: Comparison of Serratus Plane Block With Parenteral Opioid Analgesia Versus Patient Controlled Analgesia Alone in Acute Rib fracturEs
Brief Title: Serratus Plane Block With Parenteral Opioid Analgesia Versus Patient Controlled Analgesia in Rib Fractures
Acronym: COPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C&W19/007
Record Dates: First submitted 2019-04-08; First posted 2019-04-18 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Thoracic Injuries; Rib Fractures; Anaesthesia, Local; Levobupivacaine; Analgesia, Patient-Controlled; Pain
MeSH Terms: conditions — Thoracic Injuries; Rib Fractures; Agnosia; Pain | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus plane block and patient controlled analgesia (Experimental): Initial local anaesthetic bolus of 0.4 ml/kg of 0.25% levobupivacaine. Subsequent continuous local anaesthetic infusion of 0.125% levobupivacaine
  Patient controlled analgesia programmed with morphine to deliver on demand boluses of 1 mg and limited by a lockout time of 5 minutes
  Interventions: Procedure: Serratus plane block; Other: Patient controlled analgesia
- Patient controlled analgesia only (Active Comparator): Patient controlled analgesia programmed with morphine to deliver on demand boluses of 1 mg and limited by a lockout time of 5 minutes
  Interventions: Other: Patient controlled analgesia

INTERVENTIONS:
Procedure: Serratus plane block — Placement of initial local anaesthetic bolus and catheter for continuous infusion in the plane between latissimus dorsi and serratus anterior in the midaxillary line at the level of the 5th rib
  Other Names: Experimental
  Arms: Serratus plane block and patient controlled analgesia
Other: Patient controlled analgesia — Computerised pump device facilitating the patient self administration and titration as needed of morphine
  Other Names: Active comparator

SUMMARY:
In this multicentre randomised controlled trial, adult patients with isolated chest trauma and two or more unilateral rib fractures will be randomised to either serratus plane block and patient controlled analgesia or patient controlled analgesia alone. Our primary outcome is the static visual analogue scale score at one hour.

DETAILED DESCRIPTION:
Rib breaks, or fractures, can cause pain that can be very difficult to manage and can result in chest infection and death. Such pain can be managed with either systemic drugs like morphine, which are given by mouth or through the veins, or local anaesthetic techniques, which can numb the painful area. Use of systemic drugs is however limited by significant side effects and traditional local anaesthetic techniques have problems of their own. Epidural analgesia, where local anaesthetic is placed near the spine, can only be done by those with a high level of technical skill and cannot be performed in patients with spine injuries, positioning difficulties and clotting problems. Complications and side effects can be common and/or serious and include failure, fall in blood pressure, and nerve and spinal cord damage. More recently, there has been interest in a new local anaesthetic technique, serratus plane block. Serratus plane block is simple to learn and can be done without any need for repositioning of the patient. It avoids some of the complications and side effects related to other local anaesthetic techniques and is more easily looked after by nursing staff on the ward. In view of this, we are aiming to recruit 44 adults with isolated chest injury and two or more rib fractures on one side. Each patient will either receive a serratus plane block in conjunction with morphine through the veins or just morphine alone. Our main aim is to assess how bad the pain is at 1 hour, but we will also compare the pain score, morphine consumption, lung function, level of sleepiness, and the frequency of low blood pressure, nausea and vomiting and slow breathing over the first 72 hours, as well as the hospital length of stay and occurrence of lung infection within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Isolated chest trauma
* Two or more unilateral rib fractures

Exclusion Criteria:

* One unilateral rib fracture
* Bilateral rib fractures
* Flail chest
* Clavicular fractures
* Polytrauma
* Sternal fracture or injury
* Thoracic spine injury
* GCS less than 15
* Acute or chronic confusional state
* Delirium or psychiatric illness
* Chronic lung disease necessitating home nebulisers and/or oxygen
* Coagulopathy, defined as a platelet count less than 100 x 109/l , PT >15 or APTT >38
* End stage liver disease
* Severe congestive cardiac failure
* Significant renal failure, defined as a creatinine >150µmol/l
* Local infection at potential site of SBP insertion
* Pregnancy or breastfeeding
* History of chronic pain or opioid dependence
* Current chronic analgesic therapy, not to include paracetamol, NSAIDs and/or codeine
* Requirement for tracheal intubation and mechanical ventilation
* Allergy to local anaesthetics and/or opioids
* Inability to control and self-administer opioids with PCA due to confusion, learning difficulties or poor manual dexterity
* Unable to speak and/or understand English
* Patients known to clinicians to be COVID-19 positive as determined by PCR or for whom there is a clinical suspicion that they might be COVID-19 positive will be excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Static visual analogue score (0-10) at 1 hour | Measured at 1 hour
  Defined as pain score at rest

SECONDARY OUTCOMES:
Dynamic visual analogue score (0-10) | Measured at 1 hour, 24, 48 and 72 hours
  Defined as pain score on deep inspiration
Static visual analogue score (0-10) | Measured at 24, 48 and 72 hours
  Defined as pain score at rest
Morphine consumption | Measured at 24, 48 and 72 hours
  Amount of intravenous morphine consumed within each 24 hour period
Peak expiratory flow rate | Measured at 1, 24, 48 and 72 hours
  Calculated as a percentage of predicted
Level of sedation | Measured at 24, 48 and 72 hours
  Assessed using the Ramsay Sedation Scale (1-6) and a value of 2 is considered the best outcome
Incidence of hypotension | Measured at 24, 48 and 72 hours
  Defined as a systolic blood pressure less than 90 mmHg
Incidence of nausea and vomiting | Measured at 24, 48 and 72 hours
  Assessed using the Nausea-Vomiting Scale (1-4) and lower values are considered a better outcome
Incidence of respiratory depression | Measured at 24, 48 and 72 hours
  Defined as a respiratory rate of less than 12 breaths per minute
Occurence of pneumonia | Within 30 days
  Defined as occurence of in-hospital pneumonia from admission to discharge of this hospitalisation.
Hospital length of stay | Up to 6 months
  Defined as the number of days the patient stayed in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Damon Foster, Study Chair — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Sirmali M, Turut H, Topcu S, Gulhan E, Yazici U, Kaya S, Tastepe I. A comprehensive analysis of traumatic rib fractures: morbidity, mortality and management. Eur J Cardiothorac Surg. 2003 Jul;24(1):133-8. doi: 10.1016/s1010-7940(03)00256-2. PMID 12853057
- [Background] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Background] Fabricant L, Ham B, Mullins R, Mayberry J. Prolonged pain and disability are common after rib fractures. Am J Surg. 2013 May;205(5):511-5; discusssion 515-6. doi: 10.1016/j.amjsurg.2012.12.007. PMID 23592156
- [Background] Gordy S, Fabricant L, Ham B, Mullins R, Mayberry J. The contribution of rib fractures to chronic pain and disability. Am J Surg. 2014 May;207(5):659-62; discussion 662-3. doi: 10.1016/j.amjsurg.2013.12.012. Epub 2014 Jan 31. PMID 24612969
- [Background] Stawicki SP, Grossman MD, Hoey BA, Miller DL, Reed JF 3rd. Rib fractures in the elderly: a marker of injury severity. J Am Geriatr Soc. 2004 May;52(5):805-8. doi: 10.1111/j.1532-5415.2004.52223.x. PMID 15086666
- [Background] Battle CE, Hutchings H, Evans PA. Risk factors that predict mortality in patients with blunt chest wall trauma: a systematic review and meta-analysis. Injury. 2012 Jan;43(1):8-17. doi: 10.1016/j.injury.2011.01.004. Epub 2011 Jan 22. PMID 21256488
- [Background] Liman ST, Kuzucu A, Tastepe AI, Ulasan GN, Topcu S. Chest injury due to blunt trauma. Eur J Cardiothorac Surg. 2003 Mar;23(3):374-8. doi: 10.1016/s1010-7940(02)00813-8. PMID 12614809
- [Background] Clark GC, Schecter WP, Trunkey DD. Variables affecting outcome in blunt chest trauma: flail chest vs. pulmonary contusion. J Trauma. 1988 Mar;28(3):298-304. doi: 10.1097/00005373-198803000-00004. PMID 3351988
- [Background] Dehghan N, de Mestral C, McKee MD, Schemitsch EH, Nathens A. Flail chest injuries: a review of outcomes and treatment practices from the National Trauma Data Bank. J Trauma Acute Care Surg. 2014 Feb;76(2):462-8. doi: 10.1097/TA.0000000000000086. PMID 24458051
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Bayouth L, Safcsak K, Cheatham ML, Smith CP, Birrer KL, Promes JT. Early intravenous ibuprofen decreases narcotic requirement and length of stay after traumatic rib fracture. Am Surg. 2013 Nov;79(11):1207-12. PMID 24165259
- [Background] Yang Y, Young JB, Schermer CR, Utter GH. Use of ketorolac is associated with decreased pneumonia following rib fractures. Am J Surg. 2014 Apr;207(4):566-72. doi: 10.1016/j.amjsurg.2013.05.011. Epub 2013 Oct 7. PMID 24112670
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Duch P, Moller MH. Epidural analgesia in patients with traumatic rib fractures: a systematic review of randomised controlled trials. Acta Anaesthesiol Scand. 2015 Jul;59(6):698-709. doi: 10.1111/aas.12475. Epub 2015 Feb 13. PMID 25683770
- [Background] Bulger EM, Edwards T, Klotz P, Jurkovich GJ. Epidural analgesia improves outcome after multiple rib fractures. Surgery. 2004 Aug;136(2):426-30. doi: 10.1016/j.surg.2004.05.019. PMID 15300210
- [Background] Cook TM, Counsell D, Wildsmith JA; Royal College of Anaesthetists Third National Audit Project. Major complications of central neuraxial block: report on the Third National Audit Project of the Royal College of Anaesthetists. Br J Anaesth. 2009 Feb;102(2):179-90. doi: 10.1093/bja/aen360. Epub 2009 Jan 12. PMID 19139027
- [Background] Moore DC. Intercostal nerve block: spread of india ink injected to the rib's costal groove. Br J Anaesth. 1981 Apr;53(4):325-9. doi: 10.1093/bja/53.4.325. PMID 7225265
- [Background] Cheema S, Richardson J, McGurgan P. Factors affecting the spread of bupivacaine in the adult thoracic paravertebral space. Anaesthesia. 2003 Jul;58(7):684-7. doi: 10.1046/j.1365-2044.2003.03189_1.x. PMID 12886912
- [Background] Naja ZM, El-Rajab M, Al-Tannir MA, Ziade FM, Tayara K, Younes F, Lonnqvist PA. Thoracic paravertebral block: influence of the number of injections. Reg Anesth Pain Med. 2006 May-Jun;31(3):196-201. doi: 10.1016/j.rapm.2005.12.004. PMID 16701182
- [Background] Shanti CM, Carlin AM, Tyburski JG. Incidence of pneumothorax from intercostal nerve block for analgesia in rib fractures. J Trauma. 2001 Sep;51(3):536-9. doi: 10.1097/00005373-200109000-00019. PMID 11535906
- [Background] Dravid RM, Paul RE. Interpleural block - part 2. Anaesthesia. 2007 Nov;62(11):1143-53. doi: 10.1111/j.1365-2044.2007.05181.x. PMID 17924896
- [Background] Tighe SQ, Karmakar MK. Serratus plane block: do we need to learn another technique for thoracic wall blockade? Anaesthesia. 2013 Nov;68(11):1103-6. doi: 10.1111/anae.12423. Epub 2013 Sep 14. No abstract available. PMID 24032664
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Kunigo T, Murouchi T, Yamamoto S, Yamakage M. Injection Volume and Anesthetic Effect in Serratus Plane Block. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):737-740. doi: 10.1097/AAP.0000000000000649. PMID 28891826
- [Background] Mayes J, Davison E, Panahi P, Patten D, Eljelani F, Womack J, Varma M. An anatomical evaluation of the serratus anterior plane block. Anaesthesia. 2016 Sep;71(9):1064-9. doi: 10.1111/anae.13549. Epub 2016 Jul 20. PMID 27440171
- [Background] Working Party:; Association of Anaesthetists of Great Britain & Ireland; Obstetric Anaesthetists' Association; Regional Anaesthesia UK. Regional anaesthesia and patients with abnormalities of coagulation: the Association of Anaesthetists of Great Britain & Ireland The Obstetric Anaesthetists' Association Regional Anaesthesia UK. Anaesthesia. 2013 Sep;68(9):966-72. doi: 10.1111/anae.12359. Epub 2013 Aug 1. PMID 23905877
- [Background] Ochroch EA, Gottschalk A. Impact of acute pain and its management for thoracic surgical patients. Thorac Surg Clin. 2005 Feb;15(1):105-21. doi: 10.1016/j.thorsurg.2004.08.004. PMID 15707349
- [Background] Okmen K, Okmen BM. The efficacy of serratus anterior plane block in analgesia for thoracotomy: a retrospective study. J Anesth. 2017 Aug;31(4):579-585. doi: 10.1007/s00540-017-2364-9. Epub 2017 Apr 26. PMID 28447227
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192
- [Background] Lopez-Matamala B, Fajardo M, Estebanez-Montiel B, Blancas R, Alfaro P, Chana M. A new thoracic interfascial plane block as anesthesia for difficult weaning due to ribcage pain in critically ill patients. Med Intensiva. 2014 Oct;38(7):463-5. doi: 10.1016/j.medin.2013.10.005. Epub 2013 Nov 26. No abstract available. PMID 24289954
- [Background] Kunhabdulla NP, Agarwal A, Gaur A, Gautam SK, Gupta R, Agarwal A. Serratus anterior plane block for multiple rib fractures. Pain Physician. 2014 Jul-Aug;17(4):E553-5. No abstract available. PMID 25054407
- [Background] Durant E, Dixon B, Luftig J, Mantuani D, Herring A. Ultrasound-guided serratus plane block for ED rib fracture pain control. Am J Emerg Med. 2017 Jan;35(1):197.e3-197.e6. doi: 10.1016/j.ajem.2016.07.021. Epub 2016 Jul 19. No abstract available. PMID 27595172
- [Background] Fu P, Weyker PD, Webb CA. Case Report of Serratus Plane Catheter for Pain Management in a Patient With Multiple Rib Fractures and an Inferior Scapular Fracture. A A Case Rep. 2017 Mar 15;8(6):132-135. doi: 10.1213/XAA.0000000000000431. PMID 28291768